CLINICAL TRIAL: NCT01725438
Title: Clinical Validation of the ISET Method for the Non Invasive Prenatal Diagnosis of Trisomy 21 by Genetic Analysis of Circulating Trophoblastic Cells
Brief Title: Non Invasive Prenatal Diagnosis of Trisomy 21 by Genetic Analysis of Circulating Fetal Cells
Acronym: ISETTRI21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Rarecells (Industry); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM10123; P100118 (Other: AP-HP)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Trisomy 21
Keywords: Circulating Trophoblastic Cells; Non-Invasive Prenatal Diagnosis; Genetic analysis; Trisomy 21; Down's Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Noninvasive Ventilation; Noninvasive Prenatal Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnant women accepting an invasive prenatal diagnosis (Experimental): Pregnant women accepting an invasive prenatal diagnosis and a sample blood (non invasive diagnosis)
  Interventions: Other: sample blood

INTERVENTIONS:
Other: sample blood
  Other Names: Non Invasive; Prenatal Diagnosis; Trisomy 21

SUMMARY:
The objective of this project is to develop a non-invasive prenatal diagnostic test for trisomy 21 which is reliable, sensitive and cost-effective, and thus, offers an alternative to the currently employed invasive diagnostic tests amniocentesis and chorionic villus sampling.

Current prenatal screening methods (blood markers and ultrasound) for trisomy 21 (Down syndrome) detect about 90 % of cases and have a false positive rate of > 90 %. The results of these tests are expressed in risks for trisomy 21, the threshold being in France at 1/250. Women exhibiting a higher risk are offered to undergo invasive diagnostic testing, either by amniocentesis or chorionic villus sampling. However, these invasive diagnostic methods are associated with a considerable risk of miscarriage (1-3 %), and thus underline the importance to develop a safe and non-invasive prenatal diagnostic test for trisomy 21. The investigators have planned to assess the clinical impact of a non-invasive prenatal method to detect Trisomy 21 through genetic analysis of circulating trophoblastic cells.

DETAILED DESCRIPTION:
The investigators have planned and developed the following approach: fetal cells are first enriched from blood of pregnant women, between 7 and 12 weeks gestation, employing the ISET (isolation by size of epithelial tumor cells) technique. Cells presumed to be of fetal origin are microdissected and subsequently genetically analyzed, using STR markers, to verify their fetal nature. The investigators then plan to test two strategies in order to assess the number of copies of chromosome 21. The first one involves the DNA of a single fetal cell to be analyzed with CGH (comparative genomic hybridization) array. In fact, our team has already developed an application of the metaphase CGH method to single cells isolated by ISET in which we were able to demonstrate the gain of chromosome 21 DNA in single fetal cells isolated from cord blood of a fetus with Down syndrome. The second strategy will be accomplished with the use of quantitative fluorescent PCR analysis of short tandem repeats (STRs), applied to single cells. At least 5-8 highly polymorphic STR markers specific for chromosome 21 will be tested to minimize the effects of a phenomenon called allele drop out, in which one allele fails to amplify, and to maximize the number of triallelic signals for an accurate diagnosis of disomy or trisomy 21.

This survey is performed in collaboration with the Department of Gynaecology-Obstetrics - Reproductive Medicine of Antoine Béclère Hospital in Clamart. The women included in the survey will be taken a 20 ml blood sample and a cervical Pap smear before the invasive test (amniocentesis). The blood sample will be treated by the ISET method within 3 hours after collection and the filter will be stored at - 20°C. The cells obtained by Pap smear will be kept in an appropriate liquid and then treated by the ISET method in the Biochemistry Laboratory of Necker Hospital. The molecular analyses directed to the Trophoblastic cells for the NI-PND of Trisomy 21 will be performed in a blind study.

The instigators have planned to use the ISET method in a blind study including 100 cases of trisomy 21 and 300 control cases with normal caryotype. This study will allow to obtain results with sensitivity higher than 97 % and specificity higher than 99 % (IC 95 % [70-100]). The validation will be obtained by the opening of the blind study and the comparison of results obtained by the invasive method (amniocentesis) and the non-invasive method.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women older than 18 years old
* Pregnant women followed at a prenatal diagnostic centre
* Pregnant woman having a risk (> 1/250) of trisomy 21 based on the combined screening "serological tests/nuchal ultrasonography "
* Sample of blood and cervical smear obtained between the 8th and the 10th WG
* Pregnant women accepting an invasive prenatal diagnosis
* Father of the child agreeing to participate in the clinical study (accepting to give a saliva sample)
* Pregnant women beneficiary of a national insurance program
* Pregnant women and fathers signing an informed consent

Exclusion Criteria:

* Pregnant women with combined risk of trisomy 21 < 1/250
* Pregnant women non accepting the invasive prenatal diagnosis
* Pregnant women participating another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
non-invasive method of PND of Trisomy 21. | 9 months
  Clinical validation of a non-invasive method of PND of Trisomy 21.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Paterlini-Bréchot, MD, PhD, Principal Investigator — Necker Enfants Malades Hospital
Locations (1):
- Hopital de Béclère, Clamart, France

REFERENCES:
- [Background] Vona G, Sabile A, Louha M, Sitruk V, Romana S, Schutze K, Capron F, Franco D, Pazzagli M, Vekemans M, Lacour B, Brechot C, Paterlini-Brechot P. Isolation by size of epithelial tumor cells : a new method for the immunomorphological and molecular characterization of circulatingtumor cells. Am J Pathol. 2000 Jan;156(1):57-63. doi: 10.1016/S0002-9440(10)64706-2. PMID 10623654
- [Background] Vona G, Beroud C, Benachi A, Quenette A, Bonnefont JP, Romana S, Dumez Y, Lacour B, Paterlini-Brechot P. Enrichment, immunomorphological, and genetic characterization of fetal cells circulating in maternal blood. Am J Pathol. 2002 Jan;160(1):51-8. doi: 10.1016/S0002-9440(10)64348-9. PMID 11786398
- [Background] Beroud C, Karliova M, Bonnefont JP, Benachi A, Munnich A, Dumez Y, Lacour B, Paterlini-Brechot P. Prenatal diagnosis of spinal muscular atrophy by genetic analysis of circulating fetal cells. Lancet. 2003 Mar 22;361(9362):1013-4. doi: 10.1016/s0140-6736(03)12798-5. PMID 12660061
- [Background] Saker A, Benachi A, Bonnefont JP, Munnich A, Dumez Y, Lacour B, Paterlini-Brechot P. Genetic characterisation of circulating fetal cells allows non-invasive prenatal diagnosis of cystic fibrosis. Prenat Diagn. 2006 Oct;26(10):906-16. doi: 10.1002/pd.1524. PMID 16832834
- [Background] Bianchi DW, Simpson JL, Jackson LG, Elias S, Holzgreve W, Evans MI, Dukes KA, Sullivan LM, Klinger KW, Bischoff FZ, Hahn S, Johnson KL, Lewis D, Wapner RJ, de la Cruz F. Fetal gender and aneuploidy detection using fetal cells in maternal blood: analysis of NIFTY I data. National Institute of Child Health and Development Fetal Cell Isolation Study. Prenat Diagn. 2002 Jul;22(7):609-15. doi: 10.1002/pd.347. PMID 12124698